CLINICAL TRIAL: NCT02782676
Title: Clinical Investigation of the Bacterially-Derived Healon5 Ophthalmic Viscosurgical Device (OVD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VSCO-109-HLN5
Record Dates: First submitted 2016-05-23; First posted 2016-05-25 (Estimated); Results first posted 2018-05-24 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Investigational Healon5 OVD (Experimental): Subjects to receive investigational Healon5 OVD in one eye and control Healon5 in the fellow eye.
  Interventions: Device: Investigational Healon5 OVD
- Approved Healon5 OVD (Active Comparator): Subjects to receive investigational Healon5 OVD in one eye and control Healon5 in the fellow eye.
  Interventions: Device: Healon5 OVD

INTERVENTIONS:
Device: Investigational Healon5 OVD — ophthalmic viscosurgical device
  Arms: Investigational Healon5 OVD
Device: Healon5 OVD — ophthalmic viscosurgical device
  Arms: Approved Healon5 OVD

SUMMARY:
Prospective, multicenter, paired-eye, randomized, masked, clinical trial of the bacterially-derived Healon5 OVD versus the currently available Healon5 OVD control.

DETAILED DESCRIPTION:
This study will include only subjects undergoing bilateral, primary, cataract extraction and intraocular lens (IOL) implantation and who meet all of the study inclusion and exclusion criteria in both eyes. Subjects who meet the inclusion/exclusion criteria and agree to participate will be randomly assigned to receive the investigational OVD in one eye and the currently-available (i.e., commercial) OVD in the fellow eye (control). Thus, a single group of subjects will provide data for both the investigational OVD and the control OVD.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 22 years of age
* Cataracts for which extraction and posterior IOL implantation have been planned for both eyes
* Potential for postoperative best corrected distance visual acuity (BCDVA) of 20/40 Snellen or better
* Clear intraocular media, other than cataract
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Signed informed consent and HIPAA authorization

Exclusion Criteria:

* Pupil abnormalities (non-reactive, fixed pupils, or abnormally shaped pupils)
* Recent ocular trauma or ocular surgery that is not resolved/stable or may affect visual outcomes or increase risk to the subject
* Prior corneal refractive (LASIK- laser-assisted in situ keratomileusis, LASEK-laser-assisted sub-epithelial keratectomy, RK- radial keratectomy, PRK- photorefractive keratectomy, etc.) or intraocular surgery
* Corneal abnormalities such as stromal, epithelial or endothelial dystrophies that are predicted to cause visual acuity losses to a level worse than 20/40 Snellen during the study
* Subjects with diagnosed degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that are predicted to cause visual acuity losses to a level worse than 20/40 Snellen during the study.
* Conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration or tilt, such as pseudoexfoliation, trauma, or posterior capsule defects
* Use of systemic or ocular medications that may affect vision
* Prior, current, or anticipated use during the course of the 3-month study of tamsulosin or silodosin (e.g., Flomax, Flomaxtra, Rapaflo) that may, in the opinion of the investigator, confound the outcome or increase the risk to the subject (e.g., poor dilation or a lack of adequate iris structure to perform standard cataract surgery)
* Poorly-controlled diabetes
* Acute, chronic, or uncontrolled systemic or ocular disease or illness that, in the opinion of the investigator, would increase the operative risk or confound the outcome(s) of the study (e.g., immunocompromised, connective tissue disease, suspected glaucoma, glaucomatous changes in the fundus or visual field, ocular inflammation, etc.).
* Known steroid responder
* Ocular hypertension of ≥ 20 mmHg, medically-controlled ocular hypertension (regardless of IOP value ), or glaucomatous changes in the optic nerve
* Endothelial cell count (ECC) lower than 1800 cells/mm2 preoperatively (based on the lowest value of the three cell counts as taken by the Konan Specular Microscope)
* Known ocular disease or pathology that may affect visual acuity or that may be expected to require retinal laser treatment or other surgical intervention during the course of the study (macular degeneration, cystoid macular edema, diabetic retinopathy, etc.)
* Patient is pregnant, plans to become pregnant, is lactating or has another condition associated with the fluctuation of hormones that could lead to refractive changes
* Concurrent participation, or participation within 45 days prior to preoperative visit, in any other clinical trial

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kendra Hileman, PhD, Study Director — Abbott Medical Optics

IPD SHARING:
Plan to Share IPD: Yes
Serious adverse event or other adverse event data and other data as needed.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 subjects are consented but not randomized or treated in the study.
  13 subjects were randomized but did not receive study OVD in either eye.
Units Other Than Participants: Eyes
Groups:
- Investigational Healon5 OVD (Bacterially-Derived): Subject received investigational Healon5 OVD in one eye and control Healon5 in the fellow eye.
  Investigational Healon5 OVD: ophthalmic viscosurgical device
- Approved Healon5 OVD (Animal-Derived): Subjects received investigational Healon5 OVD in one eye and control Healon5 in the fellow eye.
  Healon5 OVD: ophthalmic viscosurgical device
Period: Overall Study
Arm/Group | Investigational Healon5 OVD (Bacterially-Derived) | Approved Healon5 OVD (Animal-Derived)
Started | 211; 211 Eyes | 210; 210 Eyes
Completed | 211; 211 Eyes | 209; 209 Eyes
Not Completed | 0; 0 Eyes | 1; 1 Eyes
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: 208 participants received both products, while 3 only received the Bacterially-Derived OVD and 2 only received the Animal-Derived OVD for a total of 213 paired-eye and non-paired eye subjects.
Groups:
- Subjects Received OVD (Bacterial and/or Animal-Derived): Subject received study OVD (Bacterial and/or Animal Derived) in either eye.
  (NOTE: subject numbers includes both the paired-eyes and non-paired eye participants)
Arm/Group | Subjects Received OVD (Bacterial and/or Animal-Derived)
Number analyzed (Participants) | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124
  Male | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 200
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 213

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Rates of Intraocular Pressure (IOP) Spikes 30mm of Mercury (mmHg) or Greater Measured Postoperatively
Description: The cumulative rate of IOP spikes with the bacterially-derived Healon5 will be statistically non-inferior to that with the animal-derived Healon5 control using a non-inferiority margin of 10%.
Time Frame: 3 months
Population: Results are based on paired-eye subjects included in the safety population, which differs from the total number of participant (paired + non-paired eyes)safety population used in the Participant Flow.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Healon5 OVD (Bacterially-Derived) | Approved Healon5 OVD (Animal-Derived)
Number analyzed (Participants) | 208 | 208
Participants | 17 | 13

2. Primary Outcome: Mean Percent Endothelial Cell Count (ECC) Change Preoperatively vs. Postoperatively
Description: The mean percent ECC change with the bacterially-derived Healon5 will be statistically non-inferior to that with the animal-derived Healon5 control using a non-inferiority margin of 5%.
Time Frame: 3 months
Population: Results are based on paired-eye subjects included in the safety population, which differs from the total number of participant (paired + non-paired eyes) safety population used in the Participant Flow. ECC photos were taken outside of the 3-month visit window for two subjects; therefore, the data was excluded from the analysis.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Investigational Healon5 OVD (Bacterially-Derived) | Approved Healon5 OVD (Animal-Derived)
Number analyzed (Participants) | 206 | 206
percent change | -5.55 [-6.92 to -4.17] | -6.66 [-8.06 to -5.25]

3. Secondary Outcome: Ocular Serious Adverse Events (SAE)
Description: Ocular serious and/or device related adverse event rates was be tabulated with the frequency and proportion of eyes with these events reported over time and cumulatively by OVD group.
  * in the results table denotes SAEs determined to be device-related
Time Frame: 3 months
Population: The results are consist of all subjects who had any study OVD used and with data available at the time of analysis.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Investigational Healon5 OVD (Bacterially-Derived) | Approved Healon5 OVD (Animal-Derived)
Number analyzed (Participants) | 211 | 210
Number analyzed (Eyes) | 211 | 210
Eyes
  Conjunctival Laceration | 0 | 1
  Cystoid macular edema | 0 | 1
  Elevated IOP/IOP spike (30 mmHg or greater)* | 18 | 13
  IOP spike <30 mmHg, requiring treatment* | 0 | 3
  Keratitis secondary to Sjogren's | 1 | 0
  Mild TASS | 1 | 1
  Proliferative Diabetic Retinopathy | 1 | 0
  Wound leak | 0 | 1
  Mild inflammation secondary to gout | 0 | 1
  Total eyes with no SAEs | 190 | 189

4. Secondary Outcome: Mean Change in IOP From Baseline
Description: The mean change in IOP from baseline for both OVD groups over time at the 6 hour, 1 day, 1 week, 1 month, and 3 month postoperative time points are presented.
Time Frame: 3 months
Population: Results are based on paired-eye subjects included in the safety population.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | Investigational Healon5 OVD (Bacterially-Derived) | Approved Healon5 OVD (Animal-Derived)
Number analyzed (Participants) | 208 | 208
Number analyzed (eyes) | 208 | 208
mmHg
  Change in IOP from Baseline (mmHg) at 6 hours | 5.8 (6.9) | 5.2 (5.9)
  Change in IOP from Baseline (mmHg) at 1 day | 3.9 (7.0) | 3.6 (4.9)
  Change in IOP from Baseline (mmHg) 1 week | 0.7 (3.3) | 0.9 (3.5)
  Change in IOP from Baseline (mmHg) 1 month | -0.6 (2.8) | -0.6 (2.8)
  Change in IOP from Baseline (mmHg) 3 months | -1.4 (2.6) | -1.3 (2.8)

5. Secondary Outcome: Rate of IOP Spikes 30 mmHg or Greater at 3 Month Postoperatively
Description: The rate of IOP spike 30 mmHg or greater at 6 hour, 1 day, 1 week, 1 month and 3 months postoperatively was tabulated with frequency and proportion by OVD group.
Time Frame: 3 months
Population: Results are based on paired-eye subjects included in the safety population.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Investigational Healon5 OVD (Bacterially-Derived) | Approved Healon5 OVD (Animal-Derived)
Number analyzed (Participants) | 208 | 208
Number analyzed (eyes) | 208 | 208
eyes
  6 Hours | 16 | 9
  1 Day | 4 | 5
  1 Week | 0 | 0
  1 Month | 0 | 0
  3 Months | 0 | 0

6. Secondary Outcome: Grade of Inflammation: Epithelial Edema
Description: The grades of inflammation for epithelial edema was be tabulated with frequency and proportion of eyes with each grading for each event presented over time.
Time Frame: Upto 3 months
Population: The safety population consists of all subjects who had any study OVD used and with data available at the time of analysis
  Number of eyes analyzed for Control OVD at 1 month and 3 months were less than the overall number analyzed because one subject was lost to follow up.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Investigational Healon5 OVD (Bacterially-Derived) | Approved Healon5 OVD (Animal-Derived)
Number analyzed (Participants) | 211 | 210
Number analyzed (eyes) | 211 | 210
eyes
  Epithelial Edema at 6 Hours: None (0) | 144 | 141
  Epithelial Edema at 6 Hours: Trace (+1) | 42 | 47
  Epithelial Edema at 6 Hours: Mild (+2) | 20 | 17
  Epithelial Edema at 6 Hours: Moderate (+3) | 5 | 5
  Epithelial Edema at 6 Hours: Severe (+4) | 0 | 0
  Epithelial Edema at 1 Day: None (0) | 173 | 175
  Epithelial Edema at 1 Day: Trace (+1) | 24 | 21
  Epithelial Edema at 1 Day: Mild (+2) | 10 | 11
  Epithelial Edema at 1 Day: Moderate (+3) | 3 | 2
  Epithelial Edema at 1 Day: Severe (+4) | 1 | 1
  Epithelial Edema at 1 Week: None (0) | 200 | 203
  Epithelial Edema at 1 Week: Trace (+1) | 11 | 5
  Epithelial Edema at 1 Week: Mild (+2) | 0 | 2
  Epithelial Edema at 1 Week: Moderate (+3) | 0 | 0
  Epithelial Edema at 1 Week: Severe (+4) | 0 | 0
  Epithelial Edema at 1 Month: number analyzed (Participants) | 211 | 209
  Epithelial Edema at 1 Month: number analyzed (eyes) | 211 | 209
  Epithelial Edema at 1 Month: None (0) | 210 | 208
  Epithelial Edema at 1 Month: Trace (+1) | 1 | 1
  Epithelial Edema at 1 Month: Mild (+2) | 0 | 0
  Epithelial Edema at 1 Month: Moderate (+3) | 0 | 0
  Epithelial Edema at 1 Month: Severe (+4) | 0 | 0
  Epithelial Edema at 3 Month: number analyzed (Participants) | 211 | 209
  Epithelial Edema at 3 Month: number analyzed (eyes) | 211 | 209
  Epithelial Edema at 3 Month: None (0) | 211 | 209
  Epithelial Edema at 3 Month: Trace (+1) | 0 | 0
  Epithelial Edema at 3 Month: Mild (+2) | 0 | 0
  Epithelial Edema at 3 Month: Moderate (+3) | 0 | 0
  Epithelial Edema at 3 Month: Severe (+4) | 0 | 0

7. Secondary Outcome: Grade of Inflammation: Stromal Edema
Description: The grades of inflammation for stromal edema was be tabulated with frequency and proportion of eyes with each grading for each event presented over time.
Time Frame: Upto 3 months
Population: The safety population consists of all subjects who had any study OVD used and with data available at the time of analysis
  Number of eyes analyzed for Control OVD at 1 month and 3 months were less than overall number analyzed because one subject was lost to follow up.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Investigational Healon5 OVD (Bacterially-Derived) | Approved Healon5 OVD (Animal-Derived)
Number analyzed (Participants) | 211 | 210
Number analyzed (eyes) | 211 | 210
eyes
  Stromal Edema at 6 Hours: None (0) | 178 | 173
  Stromal Edema at 6 Hours: Trace (+1) | 27 | 30
  Stromal Edema at 6 Hours: Mild (+2) | 5 | 6
  Stromal Edema at 6 Hours: Moderate (+3) | 1 | 1
  Stromal Edema at 6 Hours: Severe (+4) | 0 | 0
  Stromal Edema at 1 Day: None (0) | 184 | 182
  Stromal Edema at 1 Day: Trace (+1) | 24 | 23
  Stromal Edema at 1 Day: Mild (+2) | 3 | 4
  Stromal Edema at 1 Day: Moderate (+3) | 0 | 0
  Stromal Edema at 1 Day: Severe (+4) | 0 | 1
  Stromal Edema at 1 Week: None (0) | 207 | 206
  Stromal Edema at 1 Week: Trace (+1) | 4 | 3
  Stromal Edema at 1 Week: Mild (+2) | 0 | 1
  Stromal Edema at 1 Week: Moderate (+3) | 0 | 0
  Stromal Edema at 1 Week: Severe (+4) | 0 | 0
  Stromal Edema at 1 Month: number analyzed (Participants) | 211 | 209
  Stromal Edema at 1 Month: number analyzed (eyes) | 211 | 209
  Stromal Edema at 1 Month: None (0) | 211 | 209
  Stromal Edema at 1 Month: Trace (+1) | 0 | 0
  Stromal Edema at 1 Month: Mild (+2) | 0 | 0
  Stromal Edema at 1 Month: Moderate (+3) | 0 | 0
  Stromal Edema at 1 Month: Severe (+4) | 0 | 0
  Stromal Edema at 3 Months: number analyzed (Participants) | 211 | 209
  Stromal Edema at 3 Months: number analyzed (eyes) | 211 | 209
  Stromal Edema at 3 Months: None (0) | 211 | 209
  Stromal Edema at 3 Months: Trace (+1) | 0 | 0
  Stromal Edema at 3 Months: Mild (+2) | 0 | 0
  Stromal Edema at 3 Months: Moderate (+3) | 0 | 0
  Stromal Edema at 3 Months: Severe (+4) | 0 | 0

8. Secondary Outcome: Grade of Inflammation: Cells
Description: The grades of inflammation for cells was be tabulated with frequency and proportion of eyes with each grading for each event presented over time.
Time Frame: Upto 3 months
Population: as for outcome 6
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Investigational Healon5 OVD (Bacterially-Derived) | Approved Healon5 OVD (Animal-Derived)
Number analyzed (Participants) | 211 | 210
Number analyzed (eyes) | 211 | 210
eyes
  Cells at 6 Hours: None (0) | 27 | 22
  Cells at 6 Hours: Rare (0.5+) | 45 | 51
  Cells at 6 Hours: Trace (1+) | 116 | 105
  Cells at 6 Hours: Mild (2+) | 21 | 26
  Cells at 6 Hours: Moderate (3+) | 1 | 6
  Cells at 6 Hours: Severe (4+) | 1 | 0
  Cells at 1 Day: None (0) | 46 | 36
  Cells at 1 Day: Rare (0.5+) | 29 | 38
  Cells at 1 Day: Trace (1+) | 123 | 121
  Cells at 1 Day: Mild (2+) | 9 | 14
  Cells at 1 Day: Moderate (3+) | 4 | 1
  Cells at 1 Day: Severe (4+) | 0 | 0
  Cells at 1 Week: None (0) | 119 | 134
  Cells at 1 Week: Rare (0.5+) | 87 | 72
  Cells at 1 Week: Trace (1+) | 5 | 4
  Cells at 1 Week: Mild (2+) | 0 | 0
  Cells at 1 Week: Moderate (3+) | 0 | 0
  Cells at 1 Week: Severe (4+) | 0 | 0
  Cells at 1 Month: number analyzed (Participants) | 211 | 209
  Cells at 1 Month: number analyzed (eyes) | 211 | 209
  Cells at 1 Month: None (0) | 196 | 193
  Cells at 1 Month: Rare (0.5+) | 14 | 16
  Cells at 1 Month: Trace (1+) | 1 | 0
  Cells at 1 Month: Mild (2+) | 0 | 0
  Cells at 1 Month: Moderate (3+) | 0 | 0
  Cells at 1 Month: Severe (4+) | 0 | 0
  Cells at 3 Months: number analyzed (Participants) | 211 | 209
  Cells at 3 Months: number analyzed (eyes) | 211 | 209
  Cells at 3 Months: None (0) | 207 | 206
  Cells at 3 Months: Rare (0.5+) | 4 | 3
  Cells at 3 Months: Trace (1+) | 0 | 0
  Cells at 3 Months: Mild (2+) | 0 | 0
  Cells at 3 Months: Moderate (3+) | 0 | 0
  Cells at 3 Months: Severe (4+) | 0 | 0

9. Secondary Outcome: Grade of Inflammation: Flare
Description: The grades of inflammation for flare was be tabulated with frequency and proportion of eyes with each grading for each event presented over time.
Time Frame: Upto 3 months
Population: as for outcome 6
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Investigational Healon5 OVD (Bacterially-Derived) | Approved Healon5 OVD (Animal-Derived)
Number analyzed (Participants) | 211 | 210
Number analyzed (eyes) | 211 | 210
eyes
  Flares at 6 Hours: None (0) | 118 | 112
  Flares at 6 Hours: Faint/Trace/Mild (1+) | 93 | 91
  Flares at 6 Hours: Moderate (2+) | 0 | 7
  Flares at 1 Day: None (0) | 145 | 154
  Flares at 1 Day: Faint/Trace/Mild (1+) | 64 | 55
  Flares at 1 Day: Moderate (2+) | 2 | 1
  Flares at 1 Week: None (0) | 204 | 206
  Flares at 1 Week: Faint/Trace/Mild (1+) | 7 | 4
  Flares at 1 Week: Moderate (2+) | 0 | 0
  Flares at 1 Month: number analyzed (Participants) | 211 | 209
  Flares at 1 Month: number analyzed (eyes) | 211 | 209
  Flares at 1 Month: None (0) | 210 | 209
  Flares at 1 Month: Faint/Trace/Mild (1+) | 1 | 0
  Flares at 1 Month: Moderate (2+) | 0 | 0
  Flares at 6 Months: number analyzed (Participants) | 211 | 209
  Flares at 6 Months: number analyzed (eyes) | 211 | 209
  Flares at 6 Months: None (0) | 211 | 208
  Flares at 6 Months: Faint/Trace/Mild (1+) | 0 | 1
  Flares at 6 Months: Moderate (2+) | 0 | 0

10. Secondary Outcome: Grade of Inflammation: Anterior Synechiae
Description: The grades of inflammation for Anterior Synechiae was be tabulated with frequency and proportion of eyes with each grading for each event presented over time.
Time Frame: Upto 3 months
Population: as for outcome 6
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Investigational Healon5 OVD (Bacterially-Derived) | Approved Healon5 OVD (Animal-Derived)
Number analyzed (Participants) | 211 | 210
Number analyzed (eyes) | 211 | 210
eyes
  Anterior Synechiae at 6 Hours: None (0) | 211 | 210
  Anterior Synechiae at 6 Hours: Trace (+1) | 0 | 0
  Anterior Synechiae at 6 Hours: Mild (+2) | 0 | 0
  Anterior Synechiae at 1 Day: None (0) | 211 | 209
  Anterior Synechiae at 1 Day: Trace (+1) | 0 | 0
  Anterior Synechiae at 1 Day: Mild (+2) | 0 | 1
  Anterior Synechiae at 1 Week: None (0) | 210 | 210
  Anterior Synechiae at 1 Week: Trace (+1) | 1 | 0
  Anterior Synechiae at 1 Week: Mild (+2) | 0 | 0
  Anterior Synechiae at 1 Month: number analyzed (Participants) | 211 | 209
  Anterior Synechiae at 1 Month: number analyzed (eyes) | 211 | 209
  Anterior Synechiae at 1 Month: None (0) | 211 | 209
  Anterior Synechiae at 1 Month: Trace (+1) | 0 | 0
  Anterior Synechiae at 1 Month: Mild (+2) | 0 | 0
  Anterior Synechiae at 3 Months: number analyzed (Participants) | 211 | 209
  Anterior Synechiae at 3 Months: number analyzed (eyes) | 211 | 209
  Anterior Synechiae at 3 Months: None (0) | 211 | 209
  Anterior Synechiae at 3 Months: Trace (+1) | 0 | 0
  Anterior Synechiae at 3 Months: Mild (+2) | 0 | 0

11. Secondary Outcome: Grade of Inflammation: Posterior Synechiae
Description: The grades of inflammation for Posterior Synechiae was be tabulated with frequency and proportion of eyes with each grading for each event presented over time.
Time Frame: Upto 3 Months
Population: as for outcome 6
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Investigational Healon5 OVD (Bacterially-Derived) | Approved Healon5 OVD (Animal-Derived)
Number analyzed (Participants) | 211 | 210
Number analyzed (eyes) | 211 | 210
eyes
  Posterior Synechiae at 6 Hours: None (0) | 210 | 210
  Posterior Synechiae at 6 Hours: Trace (+1) | 1 | 0
  Posterior Synechiae at 1 Day: None (0) | 211 | 210
  Posterior Synechiae at 1 Day: Trace (+1) | 0 | 0
  Posterior Synechiae at 1 Week: None (0) | 211 | 210
  Posterior Synechiae at 1 Week: Trace (+1) | 0 | 0
  Posterior Synechiae at 1 Month: number analyzed (Participants) | 211 | 209
  Posterior Synechiae at 1 Month: number analyzed (eyes) | 211 | 209
  Posterior Synechiae at 1 Month: None (0) | 211 | 209
  Posterior Synechiae at 1 Month: Trace (+1) | 0 | 0
  Posterior Synechiae 3 Months: number analyzed (Participants) | 211 | 209
  Posterior Synechiae 3 Months: number analyzed (eyes) | 211 | 209
  Posterior Synechiae 3 Months: None (0) | 211 | 209
  Posterior Synechiae 3 Months: Trace (+1) | 0 | 0

12. Secondary Outcome: Grade of Inflammation: Fibrin Presence
Description: The grades of inflammation for Fibrin Presence was be tabulated with frequency and proportion of eyes with each grading for each event presented over time.
Time Frame: Upto 3 Months
Population: as for outcome 6
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Investigational Healon5 OVD (Bacterially-Derived) | Approved Healon5 OVD (Animal-Derived)
Number analyzed (Participants) | 211 | 210
Number analyzed (eyes) | 211 | 210
eyes
  Fibrin Presence at 6 Hours: None (0) | 210 | 210
  Fibrin Presence at 6 Hours: Trace (+1) | 0 | 0
  Fibrin Presence at 6 Hours: Mild (+2) | 1 | 0
  Fibrin Presence at 1 Day: None (0) | 210 | 209
  Fibrin Presence at 1 Day: Trace (+1) | 1 | 1
  Fibrin Presence at 1 Day: Mild (+2) | 0 | 0
  Fibrin Presence at 1 Week: None (0) | 211 | 210
  Fibrin Presence at 1 Week: Trace (+1) | 0 | 0
  Fibrin Presence at 1 Week: Mild (+2) | 0 | 0
  Fibrin Presence at 1 Month: number analyzed (Participants) | 211 | 209
  Fibrin Presence at 1 Month: number analyzed (eyes) | 211 | 209
  Fibrin Presence at 1 Month: None (0) | 210 | 209
  Fibrin Presence at 1 Month: Trace (+1) | 1 | 0
  Fibrin Presence at 1 Month: Mild (+2) | 0 | 0
  Fibrin Presence at 3 Months: number analyzed (Participants) | 211 | 209
  Fibrin Presence at 3 Months: number analyzed (eyes) | 211 | 209
  Fibrin Presence at 3 Months: None (0) | 211 | 209
  Fibrin Presence at 3 Months: Trace (+1) | 0 | 0
  Fibrin Presence at 3 Months: Mild (+2) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Investigational Healon5 OVD | Approved Healon5 OVD
All-Cause Mortality (participants affected / at risk) | 0/211 | 0/210
Serious Adverse Events (participants affected / at risk) | 24/211 | 24/210
Other Adverse Events (participants affected / at risk) | 174/211 | 173/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational Healon5 OVD (N=211) | Approved Healon5 OVD (N=210)
Elevated IOP/IOP Spike (30 mmHg or greater) (Eye disorders) | 18 | 13
IOP spike <30 mmHg, requiring treatment (Eye disorders) | 0 | 3
Conjunctival Laceration (Eye disorders) | 0 | 1
Cystoid macular edema (Eye disorders) | 0 | 1
Keratitis secondary to Sjogren's (Eye disorders) | 1 | 0
Mild TASS (toxic anterior segment syndrome) (Eye disorders) | 1 | 1
Proliferative Diabetic Retinopathy (Eye disorders) | 1 | 0
wound leak (Eye disorders) | 0 | 1
Mild inflammation secondary to gout (Eye disorders) | 0 | 1
Hospitalization: tests and observation of possible transient ischemic attack and dementia (Vascular disorders) | 1 | 1
Melanoma (Skin and subcutaneous tissue disorders) | 1 | 1
Hospitalization: penumonia and flu (Immune system disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational Healon5 OVD (N=211) | Approved Healon5 OVD (N=210)
Posterior capsule opacification (Eye disorders) | 74 | 78
Blepharitis/meibomiantis (Eye disorders) | 46 | 45
dry eye/superficial punctate keratopathy/punctate epithelialerosion/tear film insufficiency (Eye disorders) | 92 | 91
Posterior vitreous detachment (Eye disorders) | 42 | 38
Elevated IOP/ocular hypertension (Eye disorders) | 17 | 17
Posterior capsule striae/wrinkles (Eye disorders) | 52 | 52
Drusen (Eye disorders) | 16 | 17
Dermatochalasis (Eye disorders) | 15 | 17
Folds in Descemet's (Eye disorders) | 51 | 57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results.

DOCUMENTS (2):
  • Study Protocol (2016-09-21): https://cdn.clinicaltrials.gov/large-docs/76/NCT02782676/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT02782676/SAP_001.pdf